CLINICAL TRIAL: NCT03224221
Title: Apatinib Combined With Chemotherapy for Esophageal Squamous Cell Cancer After the Failure of Standard Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHAT-103
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; apatinib
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — apatinib; Fluorouracil; Platinum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib with Chemotherapy (Experimental): Apatinib with Chemotherapy(Fluorouracil and platinum)，patients will receive Apatinib at 500mg/times,oral one times daily for 28 days.the dosage of the fluorouracil and platinum need to be determined by the doctors according to the actual condition of the patients
  Interventions: Drug: Apatinib; Drug: fluorouracil and platinum
- Chemotherapy (Active Comparator): Chemotherapy (Fluorouracil and platinum)，the dosage of the fluorouracil and platinum need to be determined by the doctors according to the actual condition of the patients.
  Interventions: Drug: fluorouracil and platinum

INTERVENTIONS:
Drug: Apatinib — Patients will receive Apatinib at 500mg/times,oral one times daily for 28 days
  Arms: Apatinib with Chemotherapy
Drug: fluorouracil and platinum — the dosage of the fluorouracil and platinum need to be determined by the doctors according to the actual condition of the patients

SUMMARY:
We conduct the clinical trial to further explore the efficacy and safety of Apatinib combined with chemotherapy in treating recurrent or metastatic esophageal squamous cell carcinoma after the failure of conventional treatments.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumor and esophageal squamous cell carcinoma is the main pathological type of esophageal carcinoma in China. Treatment of recurrent or metastatic esophageal squamous cell carcinoma is usually poor. New treatments were needed. Apatinib, which was approved by CFDA (China Food and Drug Administration) for the treatment of advanced gastric cancer, is a small molecule tyrosine kinase inhibitor. It competes with intracellular VEGFR-2's ATP binding sites highly and selectively, thereby blocking downstream signaling to achieve the goal of inhibiting neovascularization in tumor tissue. We have observed in clinical practice that some patients with esophageal squamous cell carcinoma have benefited from the treatment of apatinib. So we conduct a phase II clinical trial to explore the efficacy and safety of Apatinib combined with chemotherapy (platinum and fluorouracil) in treating recurrent or metastatic esophageal squamous cell carcinoma after the failure of conventional treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female patients, age:≥18 years old.
* 2.Confirmed by histology of recurrent or metastatic esophageal squamous cell carcinoma.
* 3.Patients who undergo local or recurrent metastases after surgery and / or radiotherapy and chemotherapy,at least one measurable lesion(tumor lesions CT scan length ≥ 10 mm,lymph node lesions CT scan short diameter ≥ 15 mm,scan layer thickness is not greater than 6 mm).
* 4.The ECOG physical status score: 0 to 2.
* 5.Expected survival ≥ 3 months.
* 6.Subjects received other treatment damage have been restored, which received nitroso or mitomycin interval ≥ 6 weeks; to accept other cytotoxic drugs, radiotherapy or surgery ≥ 4 weeks, and the wound has been completely healed;
* 7.The main organs function properly:

  1. blood routine examination standards to be met (14 days without blood transfusion and blood products):

     1. HB≥90g/L;
     2. ANC≥1.5×109/L;
     3. PLT≥80×109/L;
  2. biochemical tests to meet the following criteria:

     1. TBIL<1.5×ULN;
     2. ALT and AST<2.5×ULN, and <5×ULN for patients with liver metastases
     3. Serum Cr≤1.5×ULN or endogenous creatinine clearance> 45ml/min (Cockcroft-Gault formula);
* 8.The women of childbearing age must have taken reliable contraceptive measures or have a pregnancy test (serum or urine) within 7 days prior to enrollment and have a negative result and are willing to use the appropriate method at 8 weeks after the trial and the last given test contraception.For the man, consent should be given to appropriate contraception or surgical sterilization 8 weeks after the trial and at the last time the test drug was given;
* 9.Patients should be voluntary to the trial and provide with signed informed consent

Exclusion Criteria:

* 1.Pregnant or lactating women;
* 2.Patients with high blood pressure and who can not be reduced to normal range by antihypertensive therapy (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg) with myocardial infarction or myocardial infarction, arrhythmia and grade II heart Incomplete function;
* 3.Have a significant impact on oral drug absorption factors, such as unable to swallow, chronic diarrhea and intestinal obstruction;
* 4.Coagulation dysfunction(INR>1.5 or prothrombin time (PT)>ULN + 4 seconds or APTT>1.5×ULN),with bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
* 5.with a clear gastrointestinal bleeding concerns (such as local active ulcer lesions, fecal occult blood + + above), 6 months of history of gastrointestinal bleeding;
* 6.Central nervous system metastasis with symptoms;
* 7.The investigator judged other circumstances that will affect the conduct of the study and the outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-01-23 (Estimated); Study Completion 2019-06-23 (Estimated)

PRIMARY OUTCOMES:
One-year survival rate | 12 months
  The probability of survival in one year

SECONDARY OUTCOMES:
Progress free survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Incidence of Treatment-Emergent Adverse Events | Each follow up visit, assessed up to 12 months
  Safety evaluation according to the CTCAE4.0 standard, once every 1 cycle assessment
Quality of life using EORTC QLQ C30 - scale | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Life quality evaluation using EORTC QLQ C30 - scale，once every 1 cycle assessment

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China